CLINICAL TRIAL: NCT00538616
Title: A Phase IV Single Center Cross Over Clinical Study Comparing Two Different Sedations Strategies for Mechanically Ventilated Patients With Neurological Critical Illness
Brief Title: Precedex Versus Propofol-Awakening for Reducing Brain Injury Expansion
Acronym: PrePARE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Carmelo Graffagnino (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Carmelo Graffagnino, Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00002077
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Brain Injury; Intracranial Pressure
Keywords: Brain Injury
MeSH Terms: conditions — Brain Injuries | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precedex-Propofol (Active Comparator): Patients received an infusion of precedex for six hours and then a washout and then a propofol infusion for six hours.
  Interventions: Drug: Dexmedetomidine; Drug: Propofol
- Propofol- Precedex (Active Comparator): Patients received an infusion of propofol for six hours and then a washout and then a precedex infusion for six hours.
  Interventions: Drug: Dexmedetomidine; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — in this crossover study, subjects will receive 6 hours of propofol and 6 hours of precedex (randomized crossover)
  Other Names: Precedex
Drug: Propofol — in this crossover study, subjects will receive 6 hours of propofol and 6 hours of precedex (randomized crossover)
  Other Names: Diprivan

SUMMARY:
The purpose of this study is to evaluate brain injury when two different drugs (propofol and precedex) are used to sedate patients who need a neurologic exam.

DETAILED DESCRIPTION:
The hypothesis is that a neurologic exam performed when the subject has continuous infusion of precedex will result in less brain injury (where the lactate/pyruvate ratio indicates injury) then when a neurologic exam is performed on subjects receiving propofol, because that exam requires that the propofol infusion be stopped.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of Traumatic Brain Injury (TBI), Subarachnoid Hemorrhage (SAH),Intracranial Hemorrhage (ICH), stroke
* Must require (be on) mechanical ventilation
* must require (have in place) intracranial pressure (ICP) monitoring
* must require (be receiving) continuous IV sedation

Exclusion Criteria:

* Bleeding diathesis
* Glasgow Coma Scale (GCS) < 5 with fixed pupils
* Pregnant
* elevated ICP that requires deep sedation
* pulmonary instability
* Hx of Ethanol(ETOH) abuse that requires current benzodiazepine treatment for delirium - allergy to propofol or precedex
* status epilepticus
* current neuromuscular blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Graffagnino, MD, Principal Investigator — Duke University; DaiWai M Olson, PhD RN, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects approached if they had indwelling Licox catheters and were given sedation.
Pre-assignment Details: Study started at onset of shift with 1 hour washout between crossover. One subject taken off sedation prior to enrollment because they were no longer eligible
Groups:
- Precedex-Propofol: Patients received an infusion of precedex for six hours then a washout period of one hour and then a propofol infusion for six hours.
- Propofol- Precedex: Patients received an infusion of propofol for six hours then a washout period of one hour and then a precedex infusion for six hours.
Period: Overall Study
Arm/Group | Precedex-Propofol | Propofol- Precedex
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Precedex-Propofol | Propofol- Precedex | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (5.6) | 55 (8.6) | 41.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Lactate/Pyruvate (L/P)Ratio
Description: L/P ratio was measured before during and after sedation assessment. The micromole value for each dialysate (lactate and pyruvate) was reported as well as the ratio (L/P). Elevated ratios (greater than 30) were attributed to metabolic distress (relative hypoxemia)during the course of the trial.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Precedex-Propofol | Propofol- Precedex
Number analyzed (Participants) | 5 | 3
ratio | 103.1 (249.5) | 33.8 (10.7)

ADVERSE EVENTS:
Arm/Group | Precedex-Propofol | Propofol- Precedex
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3
Other Adverse Events (participants affected / at risk) | 2/5 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precedex-Propofol (N=5) | Propofol- Precedex (N=3)
Death to initial stroke (Nervous system disorders) | 1 (1) | 0 (0) — Death was not unexpected in this case prior to subject enrollment due to severity of illness on presentation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precedex-Propofol (N=5) | Propofol- Precedex (N=3)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) — Minor bradycardia Heart Rate (HR)<60 that did not require intervention
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Onset of anemia prior to enrollment
penumonia (Infections and infestations) | 1 (1) | 0 (0) — Secondary to endotracheal intubation
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Found on 3/7/2008 Study ended on 2/23/2008

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No